CLINICAL TRIAL: NCT01984346
Title: Convergence Of Epicardial And Endocardial Radiofrequency (RF) Ablation For The Treatment Of Symptomatic Persistent AF
Brief Title: CONVERGE - Epi/Endo Ablation For Treatment of Persistent Atrial Fibrillation(AF)
Acronym: CONVERGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAL-1200; IDE Number G130084 (Other: CDRH)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial Fibrillation; Convergent Procedure; Combined Epicardial/ Endocardial Ablation; Hybrid Procedure; Radiofrequency Ablation; Arrhythmia; RF Ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Intervention Model Description: 2:1 randomized (Convergent Procedure versus standalone endocardial catheter ablation) multi-center pivotal clinical study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Convergent Procedure (Experimental): Procedure/Surgery: Convergent Procedure using EPi-Sense-AF Guided Coagulation System with Endocardial Catheter Ablation Treatment
  Interventions: Device: AtriCure EPi-Sense-AF Guided Coagulation System with VisiTrax; Device: Endocardial RF Catheter ablation using Open Irrigated-tip RF Abaltion Catheter with unidirectional or bidirectional steering
- Standalone Endocardial Catheter Ablation (Active Comparator): Procedure/Surgery: Endocardial Catheter Ablation Treatment
  Interventions: Device: Endocardial RF Catheter ablation using Open Irrigated-tip RF Abaltion Catheter with unidirectional or bidirectional steering

INTERVENTIONS:
Device: AtriCure EPi-Sense-AF Guided Coagulation System with VisiTrax — Convergent Epicardial Endocardial Ablation Procedure
  Other Names: Epicardial EPi-Sense-AF Guided Coagulation System combined with endocardial RF catheter ablation
  Arms: Convergent Procedure
Device: Endocardial RF Catheter ablation using Open Irrigated-tip RF Abaltion Catheter with unidirectional or bidirectional steering — Endocardial Catheter Ablation Procedure

SUMMARY:
This is a multi-center, open label, randomized pivotal study evaluating the safety and efficacy of the EPi-Sense-AF Guided Coagulation System for the treatment of persistent AF patients, refractory or intolerant to at least one Class I and/or III Anti Arrhythmic Drug (AAD).

DETAILED DESCRIPTION:
The objective of this randomized pivotal study is to evaluate the safety and efficacy of the AtriCure EPi-Sense®-AF Guided Coagulation System with VisiTrax® for the treatment of symptomatic persistent Atrial Fibrillation (AF) patients, refractory or intolerant to at least one Class I or Class III anti-arrhythmic drug (AAD). 153 subjects from up to 27 US and 3 OUS sites. Randomized 2:1.

The primary efficacy endpoint is success or failure to be AF/AT/AFL free absent class I and III AADs except for a previously failed or intolerant class I or III AAD with no increase in dosage following the 3-month blanking period through the 12-month post procedure follow-up visit.

The primary safety endpoint is the incidence of major adverse events (MAEs) listed in the protocol for subjects undergoing the convergent procedure for the procedural to 30-day post procedure time period.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years; < 80 years
* Left atrium < 6.0 cm
* Refractory or intolerant to one AAD (class I and/or III)
* Documentation of persistent AF
* Provided written informed consent

Exclusion Criteria:

* Patients requiring concomitant surgery
* Left ventricular ejection fraction < 40%
* Pregnant or planning to become pregnant during study
* Co-morbid medical conditions that limit one year life expectancy
* Previous cardiac surgery
* History of pericarditis
* Previous cerebrovascular accident (CVA), excluding fully resolved transient Ischemic attack (TIA)
* Patients who have active infection or sepsis
* Patients with esophageal ulcers strictures and varices
* Patients with renal dysfunction who are not on dialysis
* Patients who are contraindicated for anticoagulants
* Patients who are being treated for ventricular arrhythmias
* Patients who have had a previous left atrial catheter ablation for AF
* Patients with existing Implantable Cardioverter-Defibrillator (ICDs)
* Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a study within 30 days prior to study enrollment
* Not competent to legally represent him or herself

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2013-12; Primary Completion 2019-08 (Actual); Study Completion 2023-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David DeLurgio, MD, Principal Investigator — Emory St Joseph's Hospital
Locations (27):
- United States (25):
  - Grandview Medical Center, Birmingham, Alabama
  - Heart Center Research LLC, Huntsville, Alabama
  - Rose Medical Center / Medical Center of Aurora, Denver, Colorado
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - St. Vincent's HealthCare, Jacksonville, Florida
  - Mt Sinai Medical Center, Miami Beach, Florida
  - Palm Beach Gardens Medical Center, Palm Beach Gardens, Florida
  - Emory University - St. Joseph's Hospital, Atlanta, Georgia
  - St. Vincent Medical Group Inc., Indianapolis, Indiana
  - Cardiovascular Research Foundation of Louisiana, Baton Rouge, Louisiana
  - Lahey Clinic, Burlington, Massachusetts
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Maimonides Medical Center, Brooklyn, New York
  - Staten Island University Hospital, Staten Island, New York
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University - Vidant Medical Center, Greenville, North Carolina
  - Wake Medical Center / Cary Research Group, Raleigh, North Carolina
  - Summa Health System, Akron, Ohio
  - Riverside Hospital / OhioHealth, Columbus, Ohio
  - UPMC Pinnacle Hospitals, Harrisburg, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Austin Heart PLLC, Austin, Texas
  - STAR Clinical Trials LLC, San Antonio, Texas
  - Virginia Cardiovascular Specialists, Richmond, Virginia
- United Kingdom (2):
  - St. Bartholomew's Hospital, London
  - Guy's and St. Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gill J, Crossen KJ, Blauth C, Kerendi F, Oza SR, Magnano AR, Mostovych MA, Halkos ME, Tschopp D, Osorio J, Tabereaux P, Boedefeld W, Civello K, Ahsan S, Yap J, Billakanty S, Duff S, Costantini O, Espinal E, Kiser A, Shults C, Pederson D, Garrison J, Gilligan DM, Link MG, Kowalski M, Stees C, Sperling JS, Jacobowitz I, Yang F, Greenberg YJ, De Lurgio DB. Atrial fibrillation symptom reduction and improved quality of life following the hybrid convergent procedure: a CONVERGE trial subanalysis. Ann Cardiothorac Surg. 2024 Mar 29;13(2):155-164. doi: 10.21037/acs-2023-afm-15. Epub 2023 Aug 29. PMID 38590997
- [Derived] DeLurgio DB, Crossen KJ, Gill J, Blauth C, Oza SR, Magnano AR, Mostovych MA, Halkos ME, Tschopp DR, Kerendi F, Taigen TL, Shults CC, Shah MH, Rajendra AB, Osorio J, Silver JS, Hook BG, Gilligan DM, Calkins H. Hybrid Convergent Procedure for the Treatment of Persistent and Long-Standing Persistent Atrial Fibrillation: Results of CONVERGE Clinical Trial. Circ Arrhythm Electrophysiol. 2020 Dec;13(12):e009288. doi: 10.1161/CIRCEP.120.009288. Epub 2020 Nov 13. PMID 33185144

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruiting for the CONVERGE Study began with first site IRB approval Nov 13, 2013. Recruiting locations included physician offices, clinics and site clinical study offices.
  * The first milestone for recruiting purposes was the first 25 patients treated. This milestone was reached July 06, 2015.
  * Milestone two was hit with the attainment of 50 patients treated on September 28, 2016
  * The third milestone was the approval of the total cohort of 153 patients by the FDA on November 17, 2017.
Pre-assignment Details: 10 subjects were consented but withdrew prior to assignment to a treatment arm. 5 subjects were excluded by Investigator decision, 3 subjects withdrew consent for unkown reasons and 2 subjects withdrew based on insurance coverage considerations
Period: Overall Study
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Started (FDA full approval) | 115 (Date of full approval was 8/22/13. Date of first treated patient was 01/08/14) | 55
Treated | 102 | 51
Completed (enrollment complete 153 treated) | 98 | 50
Not Completed | 17 | 5
Not completed — Physician Decision | 4 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Enrollment Closed | 8 | 1
Not completed — Insurance Coverage | 1 | 0
Not completed — Intra-operative Exclusion | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation | Total
Number analyzed (Participants) | 102 | 51 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 23 | 69
  >=65 years | 56 | 28 | 84
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 27 | 107
  Male | 22 | 24 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 100 | 50 | 150
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 96 | 50 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: cm] — Measure done in Centimeters.
  cm | 177.7 (8.43) | 173.9 (11.64) | 176.5 (9.76)
Weight [Mean (Standard Deviation); unit: Kilograms] — Measure reported in Kilograms
  Kilograms | 104.3 (19.985) | 106.25 (23.903) | 105.0 (21.31)
BMI [Mean (Standard Deviation); unit: Kg/M2] — Measurements reported in Kg/M2
  Kg/M2 | 32.99 (5.861) | 35.11 (7.128) | 33.70 (6.37)
Smoking History [Count of Participants; unit: Participants]
  Never Smoked | 45 | 28 | 73
  Past Smoker | 48 | 20 | 68
  Current Smoker | 9 | 2 | 11
  Unknown | 0 | 1 | 1
Persistent AF [Count of Participants; unit: Participants]
  Persistent AF | 64 | 24 | 88
  Long-Standing Persistent AF | 38 | 27 | 65

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint - Number of Participants to Achieve Freedom From AF/AT/AFL.
Description: This binary primary endpoint measures number of patients to achieve freedom from AF/AT/AFL absent class I and III AADs except for previously failed or intolerant I or III AAD with no increase in dosage following the 3-month blanking period through the 12 months post procedure follow-up visit will be compared between the two treatment groups using a chi-square test using a two-sided alpha of .05 to determine if superiority of the treatment arm is attained.
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
Participants | 67 | 25
Statistical Analysis 1: Comparison: Convergent Procedure vs Standalone Endocardial Catheter Ablation; Test type: Superiority; p = 0.0472, Chi-square test — A prior threshold for statistical significance was 0.05; Mean Difference (Net) = 16.7, 95% CI 2-sided [0.1 to 33.2]

2. Primary Outcome: Primary Safety Analysis
Description: The primary safety analysis will measure the number of Major Adverse Events (MAE) collected from the start of the coagulation procedure to 30 days post procedure.
Time Frame: 30 days
Measure: Number; unit: Number of events
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
Number of events | 8 | 0

3. Secondary Outcome: Secondary Safety Endpoint - Serious Adverse Events Through 12 Months Post-procedure.
Description: The secondary safety endpoint for the study was the number of participants with serious adverse events (SAEs) in the study through the 12-months post-procedure.
Time Frame: 12 month
Population: Summary of Serious Adverse Events within 12 months occurring in >3% of the subjects in any treatment group (Safety Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
Participants
  Cardiac Disorders-Cardiac Tamponade | 4 | 0
  Cardiac Disorders- Pericardial Effusion | 4 | 0
  Cardiac Disorders- Pericarditis | 3 | 0
  Cardiac Disorders- Sinus Node Dysfunction | 0 | 2
  Cardiac Disorders-Cardiac Failure Congestive | 5 | 1
  Infections and Infestations- Pneumonia | 3 | 4
  Respiratory, Thoracic & Mediastinal Disorder- Pulmonary Edema | 3 | 0
  General Disorder and Administration Site-Chest Pain | 3 | 0
  Not applicable | 77 | 44

4. Secondary Outcome: Number of Patients With AF Burden Reduction of at Least 90% at 12 Months Compared to Baseline
Description: AF Burden Reduction of at Least 90% at 12-Months (ITT Population): The first secondary effectiveness endpoint in the fixed-sequence testing was defined as at least 90% reduction in AF burden, absent of an increased dose or new class I/III AADs, at 12 months compared to baseline.
Time Frame: 12 Months
Population: The number of subjects in the EPi- Sense group that achieved at least 90% reduction at 12 months, compared to subjects in the Catheter Ablation group.
Measure: Count of Participants; unit: Participants
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
Participants | 60 | 25

5. Secondary Outcome: AF Freedom Through 12 Months- Absent of an Increased Dose or New Class I/III AAD's.
Description: Number of patients with AF Freedom through 12 Months (ITT Population) absent of an increased dose or new class I/III AAD's
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
percentage of participants | 71 [61.7 to 79.4] | 51 [37.4 to 64.7]

6. Secondary Outcome: Number of Subjects With AF Burden Reduction of at Least 90% at 12 Months Relative to Baseline, Regardless of Class I/III AADs.
Description: Number of subjects with AF freedom through 12 months achieved in the EPi-Sense group compared to subjects in the Catheter Ablation group.
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
percentage of participants | 95 [88.8 to 99.2] | 88.6 [75.4 to 96.2]

7. Secondary Outcome: Change in Atrial Fibrillation Severity Scale (AFSS)
Description: Change was calculated as the value at 12 months minus the value at baseline. The University of Toronto's Atrial Fibrillation Severity Scale (AFSS) is a composite score of overall subject-perceived severity, global well-being, atrial fibrillation frequency, and atrial fibrillation duration. The score ranges from 3 to 30, with higher scores indicating greater atrial fibrillation burden.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
score on a scale | -11.7 (7.71) | -10.3 (7.16)

8. Secondary Outcome: Change in Quality of Life Physical Health Composite Scores Using Short Form Health Survey (SF-36)
Description: Change was calculated as the value at 12 months minus the value at baseline. The 36-Item Short Form Health Survey (SF-36) is used to determine a physical composite score based on following subscales: limitations in physical activities because of health problems; limitations in usual role activities because of physical health problems; bodily pain; vitality (energy and fatigue); and general health perceptions. The subscale scores are transformed into a range from 0 to 100, with 0=worst HRQL, 100=best HRQL. The physical component scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score, with higher scores indicating better health status.
Time Frame: 12 Months
Population: Subjects evaluated for quality of life using SF- 36 survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
score on a scale | 7.3 (10.67) | 5.7 (10.49)

9. Secondary Outcome: Quality of Life-Change in SF-36 Mental Health Composite Score Using Short Form Survey (SF-36)
Description: Change was calculated as the value at 12 months minus the value at baseline. The 36-Item Short Form Health Survey (SF-36) is used to determine a mental composite score based on the following subscales: general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; and general health perceptions. The subscale scores are transformed into a range from 0 to 100, with 0=worst HRQL, 100=best HRQL. The physical and mental component scores are constructed as a T-score with a mean of 50 and standard deviation of 10 and no minimum or maximum score, with higher scores indicating better health status.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 102 | 51
score on a scale | 5.7 (10.51) | 7.7 (12.78)

10. Secondary Outcome: Change in 6-Minute Walk Score
Description: 6 minute walk score was measured by change from baseline compared to 12-months post-procedure between the EPi-Sense and Catheter Ablation groups.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 94 | 48
Meters | 9.2 (120.59) | -12.4 (190.09)

11. Secondary Outcome: Change in Left Atrial Diameter
Description: Change in Left Atrial Diameter at 6 months from baseline.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
Number analyzed (Participants) | 99 | 51
cm | 0.1 (.62) | 1.9 (6.68)

ADVERSE EVENTS:
Time Frame: 12-month post procedure
Description: ADVERSE EVENT (AE) Any undesirable clinical occurrence or change from patient's baseline (or pre-device procedure) condition, whether it is considered device related or not.
  SERIOUS ADVERSE EVENT (SAE) Serious adverse events that are deemed device-related and/or procedure-related will be captured in the study.
  MAJOR ADVERSE EVENTS (MAE) 9 specific major adverse events defined by protocol (including death) that are device procedure related
Arm/Group | Convergent Procedure | Standalone Endocardial Catheter Ablation
All-Cause Mortality (participants affected / at risk) | 2/102 | 0/51
Serious Adverse Events (participants affected / at risk) | 97/102 | 41/51
Other Adverse Events (participants affected / at risk) | 9/102 | 0/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convergent Procedure (N=102) | Standalone Endocardial Catheter Ablation (N=51)
Cardiac Failure Congestive (Cardiac disorders) | 6 (6) | 2 (2)
Cardiac Tamponade (Cardiac disorders) | 4 (4) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 4 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Sinus Node Dysfunction (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 0 (0)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocutaneous Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal Haemorrage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary Gland Mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Pain (General disorders) | 4 (4) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Multi-Organ Disorder (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2)
Cholecystitis Infective (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 3 (3) | 1 (1)
Lobar Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 4 (4)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Staphlyococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infectiion (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional Hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedure Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toponian Increased (Investigations) | 0 (0) | 1 (1)
Fluid Overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Kaposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mestastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Cervical Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
viith Nerve Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respitory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic Respitory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Plueral Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pleuratic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cardiac Ablation (Surgical and medical procedures) | 1 (1) | 0 (0)
Colostomy Closure (Surgical and medical procedures) | 1 (1) | 0 (0)
knee Arthroplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Shoulder Arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive Emergency (Vascular disorders) | 0 (0) | 1 (1)
Jugular Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Convergent Procedure (N=102) | Standalone Endocardial Catheter Ablation (N=51)
Tamponade (Cardiac disorders) | 4 (4) | 0 (0) — Major Adverse Event-Primary Safety Endpoint Measure (Safety Population)
Excessive Bleeding (Cardiac disorders) | 2 (2) | 0 (0) — Major Adverse Event-Primary Safety Endpoint Measure (Safety Population)
Phrenic Nerve Injury (Nervous system disorders) | 1 (1) | 0 (0) — Major Adverse Event-Primary Safety Endpoint Measure (Safety Population)
Stoke (General disorders) | 1 (1) | 0 (0) — Major Adverse Event-Primary Safety Endpoint Measure (Safety Population)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0) — Major Adverse Event-Primary Safety Endpoint Measure (Safety Population)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-10-02): https://cdn.clinicaltrials.gov/large-docs/46/NCT01984346/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT01984346/SAP_001.pdf